CLINICAL TRIAL: NCT02016170
Title: Pharmacodynamic Evaluation of Switching From Prasugrel to Ticagrelor: The SWAP (SWitching Anti Platelet)-3 Study
Brief Title: Pharmacodynamic Evaluation of Switching From Prasugrel to Ticagrelor
Acronym: SWAP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWAP3
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: platelet reactivity; ticagrelor; prasugrel
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ticagrelor 180mg (Experimental): Patients on prasugrel will switch to ticagrelor with a 180mg loading dose
  Interventions: Drug: Ticagrelor 180mg
- Ticagrelor 90mg (Experimental): Patients on prasugrel will switch to ticagrelor with a 90mg maintenance dose
  Interventions: Drug: Ticagrelor 90mg
- Prasugrel 10mg (Active Comparator): Patients already on prasugrel, will maintain prasugrel
  Interventions: Drug: Prasugrel 10mg

INTERVENTIONS:
Drug: Ticagrelor 180mg — After providing written informed consent, eligible patients on maintenance prasugrel meeting inclusion and exclusion criteria will be randomized in a 1:1:1 fashion to one of the following treatment arms:
  A. Ticagrelor 180 mg loading dose (two 90mg ticagrelor tablets) followed by 90 mg BID maintenance dose for 7±2 days.
  B. Ticagrelor 90 mg (one 90mg ticagrelor tablet) followed by 90 mg BID maintenance dose for 7±2 days C. Prasugrel 10 mg once daily maintenance dose for 7±2 days
  Other Names: Brilinta
  Arms: Ticagrelor 180mg
Drug: Prasugrel 10mg — After providing written informed consent, eligible patients on maintenance prasugrel therapy meeting inclusion and exclusion criteria will be randomized in a 1:1:1 fashion to one of the following treatment arms:
  A. Ticagrelor 180 mg loading dose (two 90mg ticagrelor tablets) followed by 90 mg BID maintenance dose for 7±2 days.
  B. Ticagrelor 90 mg (one 90mg ticagrelor tablet) followed by 90 mg BID maintenance dose for 7±2 days C. Prasugrel 10 mg once daily MD for 7±2 days
  Other Names: Effient
  Arms: Prasugrel 10mg
Drug: Ticagrelor 90mg — After providing written informed consent, eligible patients on maintenance prasugrel therapy meeting inclusion and exclusion criteria will be randomized in a 1:1:1 fashion to one of the following treatment arms:
  A. Ticagrelor 180 mg loading dose (two 90mg ticagrelor tablets) followed by 90 mg BID maintenance dose for 7±2 days.
  B. Ticagrelor 90 mg (one 90mg ticagrelor tablet) followed by 90 mg BID maintenance dose for 7±2 days C. Prasugrel 10 mg once daily MD for 7±2 days
  Other Names: Brilinta
  Arms: Ticagrelor 90mg

SUMMARY:
Recently, two new oral P2Y12 antagonists have been approved for clinical use: prasugrel, a third generation thienopyridine, and ticagrelor, a first in class cyclopentyltriazolopyrimidine (CPTP). These agents have been shown to be associated with more potent platelet inhibitory effects compared with clopidogrel. In addition, both agents have shown to be superior to clopidogrel in preventing recurrent ischemic events in the setting of acute coronary syndromes (ACS). Understanding how to switch patients from prasugrel to ticagrelor is an unmet need of clinical interest. The proposed PD investigation will have a prospective, randomized, parallel design aimed to show that switching patients from prasugrel to ticagrelor provides similar levels of platelet inhibition.

DETAILED DESCRIPTION:
Dual antiplatelet therapy consisting of aspirin and a P2Y12 receptor antagonist is the cornerstone of treatment for secondary prevention of thrombotic events in patients with coronary artery disease. Recently, two new oral P2Y12 antagonists have been approved for clinical use: prasugrel, a third generation thienopyridine, and ticagrelor, a first in class cyclopentyltriazolopyrimidine (CPTP). These agents have been shown to be associated with more potent platelet inhibitory effects compared with clopidogrel. In addition, both agents have shown to be superior to clopidogrel in preventing recurrent ischemic events in the setting of acute coronary syndromes (ACS). Therefore, current guidelines recommend prasugrel or ticagrelor (as first line therapy according to European Society of Cardiology) in ACS patients undergoing percutaneous coronary intervention (PCI). Despite the broader indication for ticagrelor (also medically managed ACS) and its mortality benefit, prasugrel has a higher uptake than ticagrelor in the US market, likely due to its earlier approval. Further, implementation of prasugrel into institutional protocols, particularly for ST elevation myocardial infarction (STEMI) patients undergoing primary PCI, may also be a reason for the slow uptake of ticagrelor. However, many clinicians would indeed consider ticagrelor as the long-term treatment of choice for a variety of reasons. Therefore, understanding how to switch patients from prasugrel to ticagrelor is an unmet need of clinical interest. However, currently, there are no data on the pharmacodynamic (PD) effects of switching from prasugrel to ticagrelor. The proposed PD investigation will have a prospective, randomized, parallel design aimed to show that switching patients from prasugrel to ticagrelor provides similar levels of platelet inhibition. This study will provide insights on the PD effects of switching and will help clinicians to choose the most appropriate schema to avoid complications related to inadequate antiplatelet therapy in patients with coronary artery disease if switching from prasugrel to ticagrelor is desired.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known coronary artery disease who presented with and ACS and underwent PCI.
* Age between 18 and 74 years old.
* On therapy with low-dose aspirin (81 mg) and prasugrel 10 mg/daily for at least 14 days as per standard of care

Exclusion criteria:

* History of stroke, transient ischemic attack (TIA) or intracranial bleeding.
* Known allergies to ticagrelor.
* Weight < 60 Kg
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban).
* Treatment with IIb/IIIa glycoprotein inhibitors in the last 7 days.
* Blood dyscrasia or bleeding diathesis.
* Platelet count <80x106/mL.
* Hemoglobin <10 g/dL.
* Active bleeding.
* Hemodynamic instability.
* Creatinine Clearance <30 mL/minute.
* Known severe hepatic dysfunction.
* Patients with sick sinus syndrome (SSS) or high degree atrio-ventricular block without pacemaker protection.
* Current treatment with drugs interfering with cytochrom P450 3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromycin.
* Pregnant females.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Faz GT, Rollini F, Park Y, Cho JR, Thano E, Hu J, Kureti M, Aggarwal N, Durairaj A, Been L, Zenni MM, Guzman LA, Suryadevara S, Antoun P, Bass TA, Angiolillo DJ. Pharmacodynamic Effects of Switching From Prasugrel to Ticagrelor: Results of the Prospective, Randomized SWAP-3 Study. JACC Cardiovasc Interv. 2016 Jun 13;9(11):1089-98. doi: 10.1016/j.jcin.2016.02.039. Epub 2016 Mar 21. PMID 27013060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2014 and October 2015, a total of 150 patients on maintenance DAPT with aspirin and prasugrel were identified. Of these, 83 patients meeting study entry criteria agreed to participate and provided their written informed consent.
Pre-assignment Details: One patient was excluded after providing informed consent because of inadequate venous access. Thus a total of 82 patients were randomized.
Groups:
- Ticagrelor 180mg: Patients on prasugrel will switch to ticagrelor with a 180mg loading dose followed by 90 mg BID maintenance dose for 7±2 days.
- Ticagrelor 90mg: Patients on prasugrel will switch to ticagrelor with a 90mg maintenance dose followed by 90 mg BID maintenance dose for 7±2 days
- Prasugrel 10mg: Patients already on prasugrel, will maintain prasugrel 10 mg once daily MD for 7±2 days
Period: Overall Study
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg | Prasugrel 10mg
Started | 27 | 28 | 27
Completed | 25 | 27 | 27
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg | Prasugrel 10mg | Total
Number analyzed (Participants) | 25 | 27 | 27 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10) | 57 (7) | 57 (7) | 57 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 6 | 17
  Male | 21 | 20 | 21 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 11 | 8 | 23
  White | 21 | 16 | 19 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured as P2Y12 Reaction Units (PRU) Determined by Verify Now-P2Y12 Assay
Description: The primary hypothesis of our study was that after 1 week of randomized treatment PRU levels would be non-inferior in patients switched from prasugrel to ticagrelor (two arms combined) compared with patients remaining on prasugrel.
Time Frame: 7 days
Population: Analysis was conducted in patients who received the randomized treatment and had a valid primary end point value (PRU at 1 week).
Measure: Least Squares Mean (Standard Error); unit: PRU
Groups:
- Ticagrelor: Patients switched to ticagrelor (two arms combined) with or without a loading dose and receiving ticagrelor 90 mg bid for 7 days.
- Prasugrel: Patients already on prasugrel, will maintain prasugrel 10 mg once daily MD for 7 days
Arm/Group | Ticagrelor | Prasugrel
Number analyzed (Participants) | 52 | 27
PRU | 45 (6) | 63 (9)
Statistical Analysis 1: Comparison: Ticagrelor vs Prasugrel; Test type: Non-Inferiority or Equivalence — Non-inferiority was assessed using a 95% confidence interval (CI) of the difference in mean PRU between prasugrel and ticagrelor (two arms combined). Under the assumption of 0 difference in mean PRU between ticagrelor 90 mg bid MD and prasugrel 10 mg qd MD and a common standard deviation of 60 PRU, a sample size of 24 patients per group allowed for the 95% CI to stay within ± 45 PRU with a 90% power and alpha=0.05; Mean Difference (Final Values) = -18, 95% CI 2-sided [-41 to 5]

2. Secondary Outcome: Platelet Reactivity Index (PRI) Measured by Whole Blood Vasodilator-stimulated Phosphoprotein (VASP).
Description: The secondary hypothesis of our study was that after 1 week of randomized treatment PRI levels would be non-inferior in patients switched from prasugrel to ticagrelor (two arms combined) compared with patients remaining on prasugrel. VASP was measured by quantitative flow cytometry using commercially available labelled monoclonal antibodies.
Time Frame: 7 days
Measure: Least Squares Mean (Standard Deviation); unit: PRI
Arm/Group | Ticagrelor | Prasugrel
Number analyzed (Participants) | 52 | 27
PRI | 25 (6) | 36 (9)
Statistical Analysis 1: Comparison: Ticagrelor vs Prasugrel; Test type: Non-Inferiority or Equivalence — Non-inferiority was assessed using a 95% confidence interval (CI) of the difference in mean PRU between prasugrel and ticagrelor (two arms combined); Mean Difference (Final Values) = -11, 95% CI 2-sided [-18 to -4]

ADVERSE EVENTS:
Time Frame: 1 week
Description: The treated population comprised all patients who received any dose of study medication and was considered for analysis of safety and adverse events.
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg | Prasugrel 10mg
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 10/27 | 7/28 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 180mg (N=27) | Ticagrelor 90mg (N=28) | Prasugrel 10mg (N=27)
Angioedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 180mg (N=27) | Ticagrelor 90mg (N=28) | Prasugrel 10mg (N=27)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes